CLINICAL TRIAL: NCT04369430
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of AKST4290 in Subjects With Parkinson's Disease on Stable Dopaminergic Treatment
Brief Title: Study Assessing Efficacy and Safety of AKST4290 in Subjects With Parkinson's Disease on Stable Dopaminergic Treatment
Acronym: TEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKST4290-211
Record Dates: First submitted 2020-04-13; First posted 2020-04-30 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Parkinson's Disease; Dementia; Movement Disorder; Shaking Palsy
MeSH Terms: conditions — Parkinson Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Dementia; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AKST4290 (Experimental): Subjects will receive AKST4290, 400 mg twice daily, for 12 weeks.
  Interventions: Drug: AKST4290
- Placebo (Placebo Comparator): Subjects will receive placebo, twice daily, for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKST4290 — Oral AKST4290
  Arms: AKST4290
Drug: Placebo — Oral Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of AKST4290 in subjects with Parkinson's Disease who are currently on stable dopaminergic treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of clinically established or clinically probable PD according to MDS-PD criteria with at least 1 year of PD symptoms.
* Modified Hoehn and Yahr ≤2.5.
* Have notable motor worsening during off-medication state.
* Clear-cut improvement of motor response to levodopa medications, as assessed by the investigator.
* Must be on stable dopaminergic therapy (e.g., levodopa, dopamine agonists, monoamine oxidase inhibitors, catechol-O-methyl transferase inhibitors, amantadine), for at least 8 weeks prior to enrollment and remain on stable dose during the 12-week treatment period.
* Female subjects must not be pregnant or breastfeeding. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening. WOCBP must agree to use highly effective contraception prior to study entry. Male subjects must be willing to use a barrier method of contraception.

Key Exclusion Criteria:

* Secondary or atypical parkinsonian syndromes, for example, patients with parkinsonism from encephalitis, metabolic disorders, vascular parkinsonism, drug-induced parkinsonism, multiple system atrophy, corticobasal ganglia degeneration, progressive supranuclear palsy, Lewy body dementia.
* History of any brain surgery for PD (e.g., pallidotomy, deep brain stimulation, or fetal tissue transplant).
* Conditions affecting the peripheral or central nervous system, unless related to PD, that would affect the ability to adequately perform the MDS-UPDRS and motor assessments: i.e., severe sensory neuropathy affecting arm or leg function, or stroke affecting motor or gait function.
* Significant alcohol or drug abuse within past 2 years.
* Based on ECG reading, subjects with a risk of QT prolongation.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (22):
- United States (3):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Henry Ford Hospital West Bloomfield, West Bloomfield, Michigan
  - Movement Disorder Clinic of Oklahoma PLLC, Tulsa, Oklahoma
- Estonia (2):
  - AS Ida-Tallinna Keskhaigla / East Tallinn Central Hospital, Tallinn
  - Astra Kliinik / Astra Team Clinic, Tallinn
- Germany (8):
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Krankenhaus Agatharied GmbH, Hausham
  - Paracelsus-Elena-Klinik Kassel, Kassel
  - Universitatsklinikum Leipzig, Leipzig
  - UKGM Marburg, Marburg
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Poland (5):
  - Centrum Medyczne PRATIA/ Medical Center PRATIA, Częstochowa
  - Krakowska Akademia Neurologii/ Cracow Academy of Neurology, Krakow
  - Instytut Zdrowia Dr Boczarska-Jedynak Spolka Z Oraganiczona Odpowiedzialnoscia Spolka Komandytowa/ Institute of Health dr Boczarska-Jedynak, Oświęcim
  - Medicome SP. ZO. O./ Medicome, Oświęcim
  - Neurologiczny Nzoz Centrum Leczenia Sm Osrodek Badan Klinicznych, Plewiska
- Slovakia (4):
  - Euro-Neuro, s.r.o., Neurologická ambulancia, Bratislava
  - Nemocnica Kramáre II. Neurologická klinika LF UK a UNB /2nd Dept. Of Neurology, Comenius University Faculty of Medicine and University Hospital Bratislava, Bratislava
  - Nemocnica s poliklinikou Sv. Lukáša Galanta, a. s Neurologické oddelenie /Neurology Dpt., NsP Galanta, Galanta
  - Univerzitná nemocnica Martin Neurologická klinika/University hospital Martin, Clinic of Neurology, Martin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AKST4290 | Placebo
Started | 55 | 55
Completed | 46 | 47
Not Completed | 9 | 8
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — COVID concern, Sponsor's decision | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AKST4290 | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.07) | 64.9 (6.74) | 64.0 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 34 | 34 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 55 | 55 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 54 | 53 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Grade School | 30 | 27 | 57
  University | 14 | 19 | 33
  Masters | 9 | 9 | 18
  PhD/Medical School | 2 | 0 | 2
Baseline BMI [Mean (Standard Deviation); unit: (kg/m^2)] | 28.12 (4.986) | 27.91 (4.417) | 28.02 (4.689)
Disease Duration [Mean (Standard Deviation); unit: years] — Population: Disease duration was not captured for 3 subjects who were randomized but not treated.
  years
    number analyzed (Participants) | 52 | 55 | 107
    (all) | 5.71 (3.138) | 7.62 (5.467) | 6.69 (4.571)
Modified Hoehn and Yahr [Count of Participants; unit: Participants]
  No signs of disease | 0 | 0 | 0
  Unilateral disease | 5 | 5 | 10
  Unilateral plus axial involvement | 5 | 6 | 11
  Bilateral disease, without impairment of balance | 32 | 32 | 64
  Mild bilateral disease, with recovery on pull test | 13 | 12 | 25
Movement Disorder Society's Unified PD Rating Scale (MDS-UPDRS) Part 3 in the off-medication state [Mean (Standard Deviation); unit: score on a scale] — Sum of the corresponding items for Part 3 of the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (33 scores based on 18 questions with several right, left, or both body distribution scores) in the off-medication state. Each Parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The minimum score on the MDS-UPDRS Part 3 is 0 and the maximum is 132. Population: MDPRS Part 3 in the off-medication state was not captured for 3 subjects who were randomized but not treated.
  score on a scale
    number analyzed (Participants) | 52 | 55 | 107
    (all) | 35.2 (14.17) | 38.5 (12.44) | 36.9 (13.35)

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Function During Levodopa Withdrawal.
Description: Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part 3 Motor Examination has 33 scores based on 18 questions with several right, left, or both body distribution scores. Each Parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The minimum score on the MDS-UPDRS Part 3 is 0 and the maximum is 132.
  Outcome is the mean change from Baseline in motor function during the practically defined off-medication state, defined as at least 12 hours off levodopa, at Week 12, with lower score representing better outcome.
Time Frame: Baseline to 12 weeks
Population: Modified Intent-to-Treat/Evaluables (Subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale | -4.210 (1.1844) | -5.114 (1.1839)

2. Secondary Outcome: Safety as Assessed by the Incidence, Seriousness and Severity of Adverse Events (AEs).
Description: Incidence of treatment-emergent adverse events (TEAEs) and serious TEAEs, grouped by severity, relationship to study treatment, and AEs leading to discontinuation of study participation. Incidence was presented as number of subject with TEAEs and serious TEAEs, grouped by severity, relationship to study treatment, and AEs leading to discontinuation of study participation, throughout study duration.
Time Frame: Baseline to week 14
Population: Safety Population (all subjects who received at least one dose of the study medication). Subjects with different severity or relationship to study treatment will be counted only once at the highest grade of event.
Measure: Number; unit: participants
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 52 | 55
participants
  Subjects with any TEAEs - Severity : Mild | 12 | 17
  Subjects with any TEAEs - Severity : Moderate | 6 | 9
  Subjects with any TEAEs - Severity : Severe | 1 | 0
  Subjects with any Serious TEAEs - Severity : Mild | 0 | 0
  Subjects with any Serious TEAEs - Severity : Moderate | 0 | 3
  Subjects with any Serious TEAEs - Severity : Severe | 1 | 0
  Subjects with any TEAEs - Relationship to Study Treatment: Unrelated | 9 | 14
  Subjects with any TEAEs - Relationship to Study Treatment: Possibly Related | 10 | 11
  Subjects with any TEAEs - Relationship to Study Treatment: Definitely Related | 0 | 1
  Subjects with any Serious TEAEs - Relationship to Study Treatment: Unrelated | 1 | 3
  Subjects with any Serious TEAEs - Relationship to Study Treatment: Possibly Related | 0 | 0
  Subjects with any Serious TEAEs - Relationship to Study Treatment: Definitely Related | 0 | 3
  Subjects with any TEAEs - AEs leading to discontinuation of study participation | 2 | 2
  Subjects with any Serious TEAEs - AEs leading to discontinuation of study participation | 0 | 1

3. Secondary Outcome: Evaluation of Laboratory Changes.
Description: Incidence of of abnormalities or clinically significant changes from Baseline in laboratory test data (chemistry, hematology, coagulation, and urinalysis). Incidence was presented as number of subjects abnormal labs indicating serious condition occurred within the analysis population throughout study duration.
Time Frame: Baseline to week 14
Population: Safety Population (all subjects who received at least one dose of the study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 52 | 55
Participants
  Abnormal Blood Chemistry Labs | 18 | 12
  Abnormal Hematology Labs | 2 | 1
  Abnormal Urinalysis Labs | 0 | 0
  Abnormal Coagulation Labs | 2 | 4

4. Secondary Outcome: Evaluation of Vital Sign Changes.
Description: Incidence of abnormalities or clinically-significant changes from Baseline in Vital sign measurements (blood pressure as measured in mmHg, heart rate as measured in beats per minute, and temperature as measured in degrees Fahrenheit or Celsius). Incidence was presented as number of subjects with abnormalities or clinically-significant changes from Baseline in Vital sign measurements within the analysis group throughout study duration.
Time Frame: Baseline to week 12
Population: Safety Population (all subjects who received at least one dose of the study medication); only Abnormal, Clinically Significant incidences were reported in the Outcome Measure Data Table.
Measure: Count of Participants; unit: Participants
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 46 | 48
Participants | 0 | 2

5. Secondary Outcome: Evaluation of Electrocardiogram Changes.
Description: Incidence of abnormalities or clinically-significant changes from Baseline in 12-lead electrocardiogram (ECG) QT-interval. Incidence was presented as number of subject with ECG changes throughout study duration.
Time Frame: Baseline to week 12
Population: Safety Population (all subjects who received at least one dose of the study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 47
Participants
  Normal | 35 | 26
  Abnormal, Not Clinically Significant | 10 | 16
  Abnormal, Clinically Significant | 0 | 5

6. Secondary Outcome: The Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts 1-4, Change From Baseline During the On-medication State.
Description: The MDS-UPDRS has 4 components (details below). The rating for each item is from 0 (normal) to 4 (severe). The score for each Part is obtained from the sum of the corresponding item scores, with higher scores indicating more severe impairment.
  Part I, Non-Motor Aspects (Mentation, Behavior, and Mood) of Experiences of Daily Living (13 items), score range is 0-52.
  Part II, Motor Aspects of Experiences of Daily Living (13 items), score range is 0-52.
  Part III, Motor Examination (33 items), score range is 0-132. Part IV, Motor Complications (6 items), score range is 0-24. The outcome is the mean change from Baseline motor function during the on-medication state at Week 12, with lower value representing a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale
  MDS-UPDRS Part 1 | -0.412 (0.4581) | -0.827 (0.4581)
  MDS-UPDRS Part 2 | -0.929 (0.4552) | 0.023 (0.4552)
  MDS-UPDRS Part 3 | -1.340 (1.0729) | -1.300 (1.0728)
  MDS-UPDRS Part 4 | -0.130 (0.3129) | -0.160 (0.3129)

7. Secondary Outcome: The Montreal Cognitive Assessment (MoCA), Change From Baseline in MoCA During the On-medication State.
Description: The Montreal Cognitive Assessment (MoCA) is a neuropsychological tool that requires approximately 15 minutes to assess the following domains: attention, executive function, memory, language, visuoconstructional skills, and orientation. MoCA scores range between 0 and 30, with higher scores indicating more intact cognition.
  The MoCA is administered at Baseline and Week 12 in the on-medication state. The total score will be summarized at each scheduled time point.
  The outcome is mean change from baseline in MoCA during the on-medication state at Week 12, with higher value representing a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 43 | 44
score on a scale | 0.0 (0.23) | -0.2 (0.23)

8. Secondary Outcome: The Schwab and England Activities of Daily Living (SE-ADL) Scale, Change From Baseline in SE-ADL During the On-medication State.
Description: The SE-ADL evaluates patients' perceptions of global functional capacity and dependence. Scoring is expressed in terms of percentage, in 10 steps from 100 to 0 (100% indicates completely independent, 0% indicates bedridden with impaired vegetative functions), so that the lower the score, the worse the functional status. Scores will be summarized descriptively at each scheduled time point (i.e. n, %) by treatment group. A Generalized Estimating Equations (GEE) for alternating logistic regression (ALR) with an exchangeable working correlation structure will be employed to analyze change from baseline.
  Outcome is mean change from baseline in SE-ADL during the on-medication state at Week 12, with higher values represents a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale | 1.7 (0.91) | 1.7 (0.92)

9. Secondary Outcome: The Clinical Impression of Severity Index - PD (CISI-PD), Change From Baseline in CISI-PD During the On-medication State.
Description: The CISI-PD is a severity index formed by four items (motor signs, disability, motor complications, and cognitive status), rated 0 (not at all) to 6 (very severe or completely disabled). A total score is calculated by summing the item scores, total scores range from 0-24. The outcome is the mean change from baseline in CISI-PD during the on-medication state at Week 12, with lower score represents a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale | -0.662 (0.2867) | -0.271 (0.2867)

10. Secondary Outcome: The Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39), Change From Baseline in PDQ-39 During the On-medication State.
Description: The PDQ-39 is a patient-reported outcome of 39 questions relating to 8 key areas of health and daily activities, including both motor and non-motor symptoms. The eight dimensions include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. It is scored on a scale of 0-100 with lower scores indicating better health and high scores indicating more severe symptoms, applying to all dimensions reported in the data table.
  Outcome is the mean change from baseline in PDQ-39 during the on-medication state at Week 12, with lower score represents a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale
  Mobility | -5.021 (1.8531) | -0.744 (1.8531)
  Activities of Daily Living | -5.557 (1.6972) | -3.022 (1.6972)
  Emotional Well-Being | -7.299 (1.7185) | -4.602 (1.7184)
  Stigma | -6.372 (1.4910) | -2.602 (1.4912)
  Social Support | -3.996 (1.7285) | -0.788 (1.7285)
  Cognition | -5.415 (1.5881) | -5.693 (1.5881)
  Communication | -5.736 (1.5486) | -1.826 (1.5488)
  Bodily Discomfort | -5.660 (2.2787) | -5.594 (2.2786)
  PDQ-39 Single Index | -5.649 (1.1485) | -3.107 (1.1484)

11. Secondary Outcome: The Sheehan-Suicidality Tracking Scale (S-STS), Change From Baseline in S-STS During the On-medication State.
Description: The standard version of the S-STS is a 16-item scale that assesses the seriousness of suicidality phenomena on a Likert-type scale (0-4) ranging from "not at all" (0) to "extremely" (4), where higher scores indicate more risk of suicidality. It also assesses the frequency of key phenomena and the overall time spent in suicidality. Total score is a sum of all items; total score ranges from 0-64.
  Outcome is the mean change from baseline in S-STS during the on-medication state at Week 12, with higher score represents a worse outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
score on a scale | 0.0 (0.00) | 0.0 (0.00)

12. Secondary Outcome: 10-meter Timed Walk, Change in Baseline 10-meter Timed Walk During the on and Off-medication State
Description: The 10-meter walk test is a commonly used tool for assessing gait speed in individuals with gait limitations. Gait speed is positively correlated with the amount of community ambulation and quality of life, and it is an important measure of mobility in individuals with PD, with higher value corresponds to better mobility.
  Outcome is the mean change from baseline comfortable walking speed (gait), fast walking speed (gait), during the on and off-medication state at Week 12, with higher score represents a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 44
m/s
  Comfortable Walking Speed (Off-medication) | 0.091 (0.0326) | 0.084 (0.0329)
  Comfortable Walking Speed (On-medication) | 0.030 (0.0293) | 0.041 (0.0295)
  Fast Walking Speed (Off-medication) | 0.107 (0.0413) | 0.150 (0.0417)
  Fast Walking Speed (On-medication) | 0.041 (0.0405) | 0.075 (0.0407)

13. Secondary Outcome: Hauser 3-Day Patient Diary, Change in Baseline Mean Time Spent With and Without Troublesome Dyskinesia as Measured by the Hauser 3-Day Patient Diary
Description: The Hauser Patient Diary was developed to assess functional status over a period of time in patients with motor fluctuations and dyskinesia by recording patient motor state for half-hour intervals over a 24-hour period. The outcome is mean change of Mean Time Spent with and without troublesome dyskinesia from Baseline at Week 12.
  ON/OFF-time is time when medication is providing/not providing benefit with regard to mobility, slowness, and stiffness, respectively.
  Troublesome dyskinesia is defined as dyskinesia that interfere with function or causes meaningful discomfort. Bad time is defined as the sum of off time and on time with troublesome dyskinesia. Lower value represents a better outcome. Good time is defined as the on time without dyskinesia plus on time with non-troublesome dyskinesia. Higher value represents a better outcome.
Time Frame: Baseline to week 12
Population: Modified Intent-to-Treat/Evaluables (All subjects with nonmissing Baseline and primary endpoint data)
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 45 | 45
hours
  Mean Bad Time | -1.1 (1.06) | -1.3 (1.06)
  Mean Good time | 1.7 (1.24) | 0.4 (1.24)

ADVERSE EVENTS:
Time Frame: Baseline to Week 14
Arm/Group | AKST4290 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/52 | 3/55
Other Adverse Events (participants affected / at risk) | 8/52 | 11/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKST4290 (N=52) | Placebo (N=55)
Sudden cardiac death (General disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Neuropsychiatric syndrome (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AKST4290 (N=52) | Placebo (N=55)
Nausea (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and its employees and agents, and Principal Investigator shall not disclose to any third party or use for any purpose other than in the fulfillment of their respective obligations hereunder, any data, records or other information disclosed to Institution and Principal Investigator by Sponsor or Clinical Research Organization, or generated as a result of this Study, without the prior written consent of Sponsor (or PPD as the case may be) (hereinafter, collectively "Information").

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT04369430/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT04369430/SAP_002.pdf